CLINICAL TRIAL: NCT00882336
Title: Epidemiological Study of European Cardiovascular Risk Patients: Disease Prevention and Management in Usual Daily Practice
Brief Title: European Study of Cardiovascular Risk
Acronym: EURIKA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Other Study IDs: NIS-CEU-DUM-2008/1
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Cardiovascular Risk Factors; Hyperlipidemia; Hypertension; Diabetes; Obesity; Smoking
Keywords: Cardiovascular risk management; Hyperlipidemia; Hypertension; Diabetes; Obesity
MeSH Terms: conditions — Hyperlipidemias; Hypertension; Diabetes Mellitus; Obesity; Smoking

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients 50+ years old, with at least one additional CV risk factor (with no previous CV event or hospitalization for a CV event)

SUMMARY:
The main objective of this study is to describe the management of patients with cardiovascular risk factors in primary prevention among different European countries.

The patient's participation consists of a single study visit during a routine visit of the patient to the clinic/office.

Study variables will be measured:

* By an interview between physician and patient during the visit and/or available medical records' information: social and demographic patient characteristics, relevant family medical history, current medication.
* By questions asked to the physician: physician perception of patients' CV risk factor, guidelines adherence and cost-containment.
* By measurement performed to the patient during the visit: weight, height, BMI, waist and hip circumference will be measured.
* CV risk factors (blood parameters) will be measured by collecting available data documented within the last year in the medical records and by the collection and analyses of a blood sample during the visit.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent.
* Patients 50+ years old, with at least one additional CV risk factor (with no previous CV event or hospitalisation for a CV event) from Primary Care or hospital outpatient clinic.

Exclusion Criteria:

* Subjects who are unwilling or unable to provide informed consent
* Previous CV disease event or hospitalisation for a CV event
* Current participation in a clinical trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 50+ years old, with at least one additional CV risk factor (with no previous CV event or hospitalisation for a CV event) from Primary Care or hospital outpatient clinic.Participating investigators will belong either to PC centres or hospitals, in the proportion representing the reality on where this kind of patient is managed in each country.
Sampling Method: Probability Sample
Enrollment: 7200 (Estimated)
Dates: Start 2009-05; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterol, systolic and diastolic blood pressure, Tot. cholesterol, Non-HDL cholesterol, HDL-cholesterol, waist and hip circumference, HbA1c | Cross-sectional
Gender, age, patients with diabetes and/or hypertension (%), smoker status, family medical history. | Cross-sectional

SECONDARY OUTCOMES:
BMI, Score based 10 year CHD mortality > 5%, High Risk patients (no. and %) | Cross-sectional
Use of concomitant medication: anticoagulant, anti hypertensive, antidiabetic, lipid-lowering drugs | Cross-sectional
Biomarkers: Apo-A1, Apo-B, Hs-CRP, Creatinine, albuminuria, uric acid, glomerular filtration rate. | Cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Massó, Study Director — AstraZeneca Spain
Locations (775):
- Austria (90):
  - Research Site, Alland
  - Research Site, Bad Vöslau
  - Research Site, Baden
  - Research Site, Bierbaum am Auersbach
  - Research Site, Bludenz
  - Research Site, Deutsch Jahrndorf
  - Research Site, Feldkirch
  - Research Site, Forstau
  - Research Site, Frankenmarkt
  - Research Site, Fürstenfeld
  - Research Site, Gerasdorf bei Wien
  - Research Site, Gleisdorf
  - Research Site, Graz
  - Research Site, Graz, Geidorf
  - Research Site, Graz, Gries
  - Research Site, Graz, Strassgang
  - Research Site, Graz, Waltendorf
  - Research Site, Groß-Enzersdorf
  - Research Site, Guntramsdorf
  - Research Site, Güssing
  - Research Site, Haid
  - Research Site, Hallein
  - Research Site, Handenberg
  - Research Site, Hard, Vbg
  - Research Site, Hermagor
  - Research Site, Hohenau an der March
  - Research Site, Innsbruck
  - Research Site, Jenbach
  - Research Site, Judendorf-Strassengel
  - Research Site, Kapfenberg
  - Research Site, Kaprun
  - Research Site, Klagenfurt, Saint Martin
  - Research Site, Korneuburg
  - Research Site, KOstendorf / Sbg
  - Research Site, Kraig
  - Research Site, Krems
  - Research Site, Laab im Walde
  - Research Site, Lassee
  - Research Site, Linz, Donau
  - Research Site, Minihof Liebau
  - Research Site, Mödling
  - Research Site, Neudau
  - Research Site, Neumarkt am Wallersee
  - Research Site, Neunkirchen
  - Research Site, Neustadtl-Markt
  - Research Site, Niklasdorf
  - Research Site, Ort im Innkreis
  - Research Site, Pernitz
  - Research Site, POlfing-Brunn
  - Research Site, Pöggstall
  - Research Site, Preding
  - Research Site, Pyhra, Bez. Saint POlten
  - Research Site, Rankweil
  - Research Site, Reichenau im Mühlkreis
  - Research Site, Salzburg
  - Research Site, Sankt Leonhard am Forst
  - Research Site, Sankt Pölten
  - Research Site, Sankt Veit an der Glan
  - Research Site, Schärding Innere Stadt
  - Research Site, Seewalchen
  - Research Site, Solden
  - Research Site, Stainz
  - Research Site, Stegersbach
  - Research Site, Steinakirchen am Forst
  - Research Site, Steyr
  - Research Site, Straning
  - Research Site, Tulfes
  - Research Site, Vienna
  - Research Site, Villach-Innere Stadt
  - Research Site, Vöcklabruck
  - Research Site, Waidhofen an der Thaya
  - Research Site, Waizenkirchen
  - Research Site, Weilbach, OO
  - Research Site, Wels
  - Research Site, Wien, Alsergrund
  - Research Site, Wien, DObling
  - Research Site, Wien, Donaustadt
  - Research Site, Wien, Floridsdorf
  - Research Site, Wien, Hernals
  - Research Site, Wien, Innere Stadt
  - Research Site, Wien, Josefstadt
  - Research Site, Wien, Landstrasse
  - Research Site, Wien, Leopoldstadt
  - Research Site, Wien, Mariahilf
  - Research Site, Wien, Meidling
  - Research Site, Wien, Neubau
  - Research Site, Wien, Ottakring
  - Research Site, Wien, Penzing
  - Research Site, Wiener Neustadt
  - Research Site, Ziersdorf
- Belgium (69):
  - Research Site, Aalst
  - Research Site, Aalter
  - Research Site, Anthée
  - Research Site, Ath
  - Research Site, Beauvechain
  - Research Site, Bellaire
  - Research Site, Berchem (antwerpen)
  - Research Site, Braine-le-Comte
  - Research Site, Brakel
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Céroux-Mousty
  - Research Site, Champion
  - Research Site, Chimay
  - Research Site, Cul-des-Sarts
  - Research Site, Deurne (antwerpen)
  - Research Site, Eeklo
  - Research Site, Erpe
  - Research Site, Forest
  - Research Site, Geraardsbergen
  - Research Site, Ghent
  - Research Site, Gooik
  - Research Site, Gosselies
  - Research Site, Ham-sur-Heure
  - Research Site, Hasselt
  - Research Site, Herentals
  - Research Site, Jambes (namur)
  - Research Site, Kapelle-op-den-Bos
  - Research Site, Kortrijk
  - Research Site, Kortrijk-Dutsel
  - Research Site, Kruishoutem
  - Research Site, Leignon
  - Research Site, Leuven
  - Research Site, Liernu
  - Research Site, Linkebeek
  - Research Site, Lummen
  - Research Site, Maasmechelen
  - Research Site, Maillen
  - Research Site, Mol
  - Research Site, Molenstede
  - Research Site, Moorsel
  - Research Site, Neupré
  - Research Site, Oosteeklo
  - Research Site, Ottignies
  - Research Site, Oudenaarde
  - Research Site, Robertville
  - Research Site, Roeselare
  - Research Site, Sambreville
  - Research Site, Sint-Andries
  - Research Site, Sint-Niklaas
  - Research Site, Sint-Truiden
  - Research Site, St-maria-oudenhove (zot.)
  - Research Site, Strépy-Bracquegnies
  - Research Site, Thieusies
  - Research Site, Tongeren
  - Research Site, Vaux-sous-Chèvremont
  - Research Site, Velm
  - Research Site, Verviers
  - Research Site, Veurne
  - Research Site, Villers-la-Ville
  - Research Site, Vivegnis
  - Research Site, Vorst (kempen)
  - Research Site, Walem
  - Research Site, Wavre
  - Research Site, Westouter
  - Research Site, Wetteren
  - Research Site, Wilrijk (antwerpen)
  - Research Site, Zemst
  - Research Site, Zonhoven
- France (96):
  - Research Site, Agen
  - Research Site, Aillas
  - Research Site, Aix-en-Provence
  - Research Site, Alès
  - Research Site, Annonay
  - Research Site, Anzin
  - Research Site, Arcachon
  - Research Site, Arces-Dilo
  - Research Site, Argancy
  - Research Site, Argenton-lÉglise
  - Research Site, Aucamville
  - Research Site, Aulnois-sur-Seille
  - Research Site, Auzeville-Tolosane
  - Research Site, Bagnols-en-Forêt
  - Research Site, Baulon
  - Research Site, Beausoleil
  - Research Site, Besançon
  - Research Site, Bourgoin
  - Research Site, Branne
  - Research Site, Brive-la-Gaillarde
  - Research Site, Bron
  - Research Site, Cagnes-sur-Mer
  - Research Site, Capdenac-Gare
  - Research Site, Castelnaudary
  - Research Site, Chambéry
  - Research Site, Chantilly
  - Research Site, Clermont-Ferrand
  - Research Site, Colombes
  - Research Site, Conflans STE Honorine
  - Research Site, Courpière
  - Research Site, Ennery
  - Research Site, Escaudain
  - Research Site, Fontenay-sous-Bois
  - Research Site, Gournay-en-Bray
  - Research Site, Gray
  - Research Site, Grenoble
  - Research Site, Grignols
  - Research Site, Hesdin
  - Research Site, Hyères
  - Research Site, Kunheim
  - Research Site, La Baule-Escoublac
  - Research Site, La Ferté-Saint-Aubin
  - Research Site, La Rivière-Saint-Sauveur
  - Research Site, Labergement STE Marie
  - Research Site, Le Ban Saint-Martin
  - Research Site, Les Milles
  - Research Site, Lourmarin
  - Research Site, Lyon
  - Research Site, Maizières-lès-Metz
  - Research Site, Marckolsheim
  - Research Site, Marseille
  - Research Site, Mauléon-Licharre
  - Research Site, Mauriac
  - Research Site, Mayet
  - Research Site, Meaux
  - Research Site, Metz-Tessy
  - Research Site, Méry-sur-Seine
  - Research Site, Montpellier
  - Research Site, Montreuil
  - Research Site, Mornas
  - Research Site, Nice
  - Research Site, Orange
  - Research Site, Paris
  - Research Site, Pertuis
  - Research Site, Pessac
  - Research Site, Ploeren
  - Research Site, Poissy
  - Research Site, Quimper
  - Research Site, Reims
  - Research Site, Riedisheim
  - Research Site, Rieumes
  - Research Site, Romorantin-Lanthenay
  - Research Site, Rougegoutte
  - Research Site, Rueil-Malmaison
  - Research Site, Saint Maximin LA STE Baume
  - Research Site, Saint-Aulaire
  - Research Site, Saint-Avold
  - Research Site, Saint-Guénolé
  - Research Site, Saint-Michel-Chef-Chef
  - Research Site, Saint-Omer
  - Research Site, Salles-sur-l'Hers
  - Research Site, Schweighouse-sur-Moder
  - Research Site, Sète
  - Research Site, Soissons
  - Research Site, STE MERE Eglise
  - Research Site, Toulon
  - Research Site, Tours
  - Research Site, Vélizy-Villacoublay
  - Research Site, Vidauban
  - Research Site, Vigoulet
  - Research Site, Villenave-d'Ornon
  - Research Site, Villepinte
  - Research Site, Vincennes
  - Research Site, Wingles
  - Research Site, Woippy
  - Research Site, Yerres
- Germany (55):
  - Research Site, Afritz
  - Research Site, Augsburg , Bay
  - Research Site, Bad Bentheim
  - Research Site, Bad Bocklet
  - Research Site, Bad Driburg
  - Research Site, Bad Harzburg
  - Research Site, Bad Schönborn
  - Research Site, Bad Wildbad
  - Research Site, Berlin
  - Research Site, Bernkastel-Kues
  - Research Site, Bietigheim-Bissingen
  - Research Site, Brilon
  - Research Site, BurgstAdt , Sachs
  - Research Site, Dippoldiswalde
  - Research Site, Dresden
  - Research Site, Duisburg
  - Research Site, Düsseldorf
  - Research Site, Eisenhüttenstadt
  - Research Site, Eppelheim , Baden
  - Research Site, Erlangen
  - Research Site, Erligheim
  - Research Site, Feucht
  - Research Site, Fischen I. AllgAu
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Genthin
  - Research Site, Gunzenhausen Am AltmUhlsee
  - Research Site, Hamburg
  - Research Site, Hildesheim
  - Research Site, Kaiserslautern
  - Research Site, Karlsruhe , Baden
  - Research Site, Laaber , Oberpf
  - Research Site, Langen B Bremerhaven
  - Research Site, Leverkusen
  - Research Site, Ludwigshafen am Rhein
  - Research Site, Magdeburg
  - Research Site, Neunkirchen , Saar
  - Research Site, NUrnberg , Mittelfr
  - Research Site, Offenbach
  - Research Site, Randersacker
  - Research Site, Riesa
  - Research Site, Rotenburg A. D. Fulda
  - Research Site, Scheinfeld
  - Research Site, Schongau
  - Research Site, Siegen
  - Research Site, Simmern
  - Research Site, Singen (Hohentwiel)
  - Research Site, Solingen
  - Research Site, Spremberg , NL
  - Research Site, Steinbach am Taunus
  - Research Site, Ulm , Donau
  - Research Site, Wasserburg A. Inn
  - Research Site, Wegberg
  - Research Site, Wiesbaden
  - Research Site, Würzburg
- Greece (35):
  - Research Site, Agia Marina
  - Research Site, Agrinio
  - Research Site, Alexandroupoli
  - Research Site, Amfissa
  - Research Site, Argos
  - Research Site, Argostoli
  - Research Site, Arta
  - Research Site, Athens
  - Research Site, Corinth
  - Research Site, Euvoia
  - Research Site, Grevená
  - Research Site, Halkida
  - Research Site, Heraklion-crete
  - Research Site, Igoumenitsa
  - Research Site, Ioannina
  - Research Site, Kalambaka
  - Research Site, Karditsa
  - Research Site, Katerini
  - Research Site, Kavala
  - Research Site, Kilkis
  - Research Site, Lakonia
  - Research Site, Larissa
  - Research Site, Lehaina
  - Research Site, Leptokaryá
  - Research Site, Naupaktos
  - Research Site, Pátrai
  - Research Site, Porto Rafti
  - Research Site, Stilís
  - Research Site, Stoúpa
  - Research Site, Thebes
  - Research Site, Thessaloniki
  - Research Site, Trikala
  - Research Site, Véroia
  - Research Site, Volos
  - Research Site, Xánthi
- Norway (63):
  - Research Site, Arendal
  - Research Site, Ågotnes
  - Research Site, Ålesund
  - Research Site, Ås
  - Research Site, Bergen
  - Research Site, Birtavarre
  - Research Site, Bjerkvik
  - Research Site, Bodø
  - Research Site, Brattvåg
  - Research Site, Drammen
  - Research Site, Elverum
  - Research Site, Fevik
  - Research Site, Flatanger
  - Research Site, Flekkefjord
  - Research Site, Frøland
  - Research Site, Grimstad
  - Research Site, Hafrsfjord
  - Research Site, Hallingby
  - Research Site, Hamar
  - Research Site, Harstad
  - Research Site, Hatlestrand
  - Research Site, Hof
  - Research Site, Holmestrand
  - Research Site, Hovik
  - Research Site, Hurdal
  - Research Site, Jevnaker
  - Research Site, Jørpeland
  - Research Site, Kapp
  - Research Site, Karlshus
  - Research Site, Kjøpsvik
  - Research Site, Kolvereid
  - Research Site, Kristiansand
  - Research Site, Kristiansund N
  - Research Site, Larvik
  - Research Site, Levanger
  - Research Site, Lundamo
  - Research Site, Mandal
  - Research Site, Misvær
  - Research Site, Mjøndalen
  - Research Site, Namsos
  - Research Site, Nesoddtangen
  - Research Site, Nttery
  - Research Site, Oslo
  - Research Site, Rådal
  - Research Site, Råholt
  - Research Site, Rena
  - Research Site, Romedal
  - Research Site, Rykkin
  - Research Site, Sande I Vestfo
  - Research Site, Sandefjord
  - Research Site, Sandnes
  - Research Site, Sannidal
  - Research Site, Sarpsborg
  - Research Site, Sellebakk
  - Research Site, Skien
  - Research Site, Snarya
  - Research Site, Sola
  - Research Site, Srumsand
  - Research Site, Stavanger
  - Research Site, Støren
  - Research Site, Tynset
  - Research Site, Våler
  - Research Site, Vestskogen
- Russia (3):
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Spain (91):
  - Research Site, A Coruña
  - Research Site, Abadin (casco Urbano) - LUGO
  - Research Site, Aceuchal - Badajoz
  - Research Site, Ademuz
  - Research Site, Albacete
  - Research Site, Alhaurin EL Grande-malaga
  - Research Site, Alicante
  - Research Site, Arzua-a Coruna
  - Research Site, AS Pontes - A Coruna
  - Research Site, Aviles - Asturias
  - Research Site, Ávila
  - Research Site, Barruelo de Santullan - Palencia
  - Research Site, BEAS de Segura - JAEN
  - Research Site, Begonte - LUGO
  - Research Site, Bilbao - Vizcaya
  - Research Site, Blanca - Murcia
  - Research Site, Boadilla DEL Monte - Madrid
  - Research Site, Bohonal de IBOR - C�ceres
  - Research Site, Bonavista - Tarragona
  - Research Site, Calpe- Alicante
  - Research Site, Castelldefels - Barcelona
  - Research Site, Castellon
  - Research Site, Ceuta
  - Research Site, Cieza - Murcia
  - Research Site, Ciudad Real
  - Research Site, Cornella de Llobregat - Barcelona
  - Research Site, Cuenca
  - Research Site, Daimiel - Ciudad REAL
  - Research Site, Eivissa - Illes Balears
  - Research Site, EL PRAT de Llobregat - Barcelona
  - Research Site, Elda-alicante
  - Research Site, Figueres - Girona
  - Research Site, Granada
  - Research Site, Guenes - Vizcaya
  - Research Site, Huelma - JAEN
  - Research Site, Huelva
  - Research Site, Huesca
  - Research Site, Jaén
  - Research Site, l'Alfàs del Pi
  - Research Site, L'hospitalet de Llobregat - Barcelona
  - Research Site, LA Linea de LA Concepcion - Cadiz
  - Research Site, LA Nucia-alicante
  - Research Site, LA ROCA DEL Vall�s - Barcelona
  - Research Site, LA Victoria -santa CRUZ de Tenerife
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Leganes - Madrid
  - Research Site, León
  - Research Site, LEPE - Huelva
  - Research Site, Lerma - Burgos
  - Research Site, Llica D'amunt - Barcelona
  - Research Site, Luceni - Zaragoza
  - Research Site, Madrid
  - Research Site, Majadahonda - Madrid
  - Research Site, Manzanares - Ciudad REAL
  - Research Site, Mataro - Barcelona
  - Research Site, Málaga
  - Research Site, Medina de Ríoseco
  - Research Site, Mombeltran - Avila
  - Research Site, Moron de LA Frontera - Sevilla
  - Research Site, Mostoles - Madrid
  - Research Site, Murias (mieres) - Asturias
  - Research Site, Navarres - Valencia
  - Research Site, Olite-navarra
  - Research Site, Ourense
  - Research Site, Palma de Mallorca - Illes Balears
  - Research Site, Pamplona-navarra
  - Research Site, Petrer - Alicante
  - Research Site, Redondela - Pontevedra
  - Research Site, Ronda-malaga
  - Research Site, SAN Bartolome - Orihuela - Alicante
  - Research Site, SAN Sebasti�n
  - Research Site, Santa CRUZ de Mudela - Ciudad REAL
  - Research Site, Santiago de Compostela - A Coruna
  - Research Site, Segorbe - Castellon
  - Research Site, Seville
  - Research Site, Soria
  - Research Site, Soutomaior - Pontevedra
  - Research Site, Tarragona
  - Research Site, Terrassa - Barcelona
  - Research Site, Tolosa-guipuzcoa
  - Research Site, Torrejon de Ardoz - Madrid
  - Research Site, TOSA de MAR - Girona
  - Research Site, Tudela - Navarra
  - Research Site, Valdemoro - Madrid
  - Research Site, Valencia
  - Research Site, Valladolid
  - Research Site, VIGO - Pontevedra
  - Research Site, Vilagarcia-pontevedra
  - Research Site, Vilassar de MAR- Barcelona
  - Research Site, Villaseca de LA Sagra - Toledo
  - Research Site, Zaragoza
- Sweden (53):
  - Research Site, Ängelholm
  - Research Site, Åtvidaberg
  - Research Site, Bjärred
  - Research Site, Boden
  - Research Site, Bollnäs
  - Research Site, Borlänge
  - Research Site, Dalby
  - Research Site, Enköping
  - Research Site, Eskilstuna
  - Research Site, Gävle
  - Research Site, Gothenburg
  - Research Site, Handen
  - Research Site, Helsingborg
  - Research Site, Höör
  - Research Site, Huddinge
  - Research Site, Hudiksvall
  - Research Site, Jarfalla
  - Research Site, Jönköping
  - Research Site, Karlskoga
  - Research Site, Karlstad
  - Research Site, Kil
  - Research Site, Kiruna
  - Research Site, Kristianstad
  - Research Site, Kungälv
  - Research Site, Limhamn
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Mora
  - Research Site, Norrköping
  - Research Site, Nyköping
  - Research Site, Nynäshamn
  - Research Site, Örebro
  - Research Site, Örnsköldsvik
  - Research Site, Österbybruk
  - Research Site, Östhammar
  - Research Site, Sala
  - Research Site, Sävedalen
  - Research Site, Skene
  - Research Site, Söderhamn
  - Research Site, Stockholm
  - Research Site, Sundbyberg
  - Research Site, Sunne
  - Research Site, Trelleborg
  - Research Site, Trollhättan
  - Research Site, Tullinge
  - Research Site, Tyreso
  - Research Site, Uppsala
  - Research Site, Varberg
  - Research Site, Vaxjo
  - Research Site, Värnamo
  - Research Site, Västerås
  - Research Site, Vimmerby
- Switzerland (77):
  - Research Site, Aarau
  - Research Site, Alle
  - Research Site, Allschwil
  - Research Site, Arbedo
  - Research Site, Baden
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Bernex
  - Research Site, Biel/Bienne
  - Research Site, Bironico
  - Research Site, Bi�re
  - Research Site, Bremgarten
  - Research Site, Burgdorf
  - Research Site, Cheseaux-sur-Lau
  - Research Site, Chur
  - Research Site, Ch�ne-Bourg
  - Research Site, Davos Platz
  - Research Site, Delémont
  - Research Site, Diegten
  - Research Site, Ebmatingen
  - Research Site, Egg
  - Research Site, Elsau-Räterschen / Räterschen
  - Research Site, Épalinges
  - Research Site, Fleurier
  - Research Site, Fribourg
  - Research Site, Frick
  - Research Site, Fully
  - Research Site, Genolier
  - Research Site, Gen�ve
  - Research Site, Gland
  - Research Site, Glattbrug
  - Research Site, Grono
  - Research Site, Ilanz
  - Research Site, Interlaken
  - Research Site, Kerns
  - Research Site, Küsnacht
  - Research Site, Lausanne
  - Research Site, Le Noirmont
  - Research Site, Le Sentier
  - Research Site, Les Acacias
  - Research Site, Leysin
  - Research Site, Locarno
  - Research Site, Lonay
  - Research Site, Lucerne
  - Research Site, Lugano
  - Research Site, Luthern Dorf
  - Research Site, Montreux
  - Research Site, Moutier
  - Research Site, Neerach
  - Research Site, Nyon
  - Research Site, Oberweningen
  - Research Site, Onex
  - Research Site, Orbe
  - Research Site, Ostermundigen
  - Research Site, Pfeffingen
  - Research Site, Porrentruy
  - Research Site, Posieux
  - Research Site, Rapperswil
  - Research Site, Reinach
  - Research Site, Rothenburg
  - Research Site, Saint-Imier
  - Research Site, Sankt Gallen
  - Research Site, Schänis
  - Research Site, Schiers
  - Research Site, Sierre
  - Research Site, Thun
  - Research Site, Unterägeri
  - Research Site, Urnäsch
  - Research Site, Vevey
  - Research Site, Villeneuve
  - Research Site, Weggis
  - Research Site, Weisslingen
  - Research Site, Winterthur
  - Research Site, Worb
  - Research Site, Zollikofen
  - Research Site, Zurich
  - Research Site, Zweisimmen
- Turkey (Türkiye) (53):
  - Research Site, Adıyaman
  - Research Site, Altındağ
  - Research Site, Anamur
  - Research Site, Ankara
  - Research Site, Avcılar
  - Research Site, Bafra
  - Research Site, Buca
  - Research Site, Buharkent
  - Research Site, Buyukcekm
  - Research Site, Çankaya
  - Research Site, Çeltikçi
  - Research Site, Çine
  - Research Site, Çorum
  - Research Site, Didim
  - Research Site, Fatih
  - Research Site, Gebze
  - Research Site, Gölhisar
  - Research Site, Havran
  - Research Site, Havsa
  - Research Site, Heraclea
  - Research Site, Kadıköy
  - Research Site, Kağızman
  - Research Site, Karasu
  - Research Site, Kargı
  - Research Site, Keles
  - Research Site, Kilis
  - Research Site, Kocasinan
  - Research Site, Kürtün
  - Research Site, Kırklareli
  - Research Site, Lefkose
  - Research Site, Magosa
  - Research Site, Manavgat
  - Research Site, Manisa
  - Research Site, Melikgazi
  - Research Site, Menemen
  - Research Site, Mersin
  - Research Site, Nilufer
  - Research Site, Ondokuzmayıs
  - Research Site, Osmangazi
  - Research Site, Pendik/ Kaynarca
  - Research Site, Reşadiye
  - Research Site, Rize
  - Research Site, Sanliurfa
  - Research Site, Sinop
  - Research Site, Sivas
  - Research Site, Şişli
  - Research Site, Tarsus
  - Research Site, Tepebaşı
  - Research Site, Türkoğlu
  - Research Site, Van
  - Research Site, Yeşilköy
  - Research Site, Yozgat
  - Research Site, Yüksekova
- United Kingdom (90):
  - Research Site, Amersham
  - Research Site, Atherstone
  - Research Site, Axbridge
  - Research Site, Aylesbury
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Bordon
  - Research Site, Borehamwood
  - Research Site, Bradford-on-Avon
  - Research Site, Bridport
  - Research Site, Bristol
  - Research Site, Brough
  - Research Site, Bude
  - Research Site, Burntwood
  - Research Site, Calne
  - Research Site, Camberley
  - Research Site, Camborne
  - Research Site, Cambridge
  - Research Site, Chippenham
  - Research Site, Chislehurst
  - Research Site, Cleethorpes
  - Research Site, Cowbridge
  - Research Site, Cranbrook
  - Research Site, Crawley
  - Research Site, Croydon
  - Research Site, Cumbernauld
  - Research Site, Dawlish
  - Research Site, Doncaster
  - Research Site, Dumfries
  - Research Site, Dunfermline
  - Research Site, Edgware
  - Research Site, Edinburgh
  - Research Site, Ely
  - Research Site, Enfield
  - Research Site, Epsom
  - Research Site, Exeter
  - Research Site, Falmouth
  - Research Site, Frome
  - Research Site, Gillingham
  - Research Site, Glasgow
  - Research Site, Great Missenden
  - Research Site, Harrow
  - Research Site, Hayes
  - Research Site, Horsham
  - Research Site, Huddersfield
  - Research Site, Ilford
  - Research Site, Ipswich
  - Research Site, Isle of Arran
  - Research Site, Isle of Man
  - Research Site, Jersey
  - Research Site, Kettering
  - Research Site, Leatherhead
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, Leven
  - Research Site, Lincoln
  - Research Site, London
  - Research Site, Louth
  - Research Site, Manchester
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Midhurst
  - Research Site, Milton Keynes
  - Research Site, Mountain Ash
  - Research Site, Neath
  - Research Site, Newport
  - Research Site, Newtownabbey
  - Research Site, Newtownards
  - Research Site, Normanton
  - Research Site, Northampton
  - Research Site, Norwich
  - Research Site, Nottingham
  - Research Site, Oxford
  - Research Site, Paignton
  - Research Site, Peterhead
  - Research Site, Plymouth
  - Research Site, Preston
  - Research Site, Reading
  - Research Site, Rochdale
  - Research Site, Ruislip
  - Research Site, Saint Leonards-on-Sea
  - Research Site, Seaton
  - Research Site, Sheffield
  - Research Site, Skelmersdale
  - Research Site, Smethwick
  - Research Site, Stafford
  - Research Site, Stratford-upon-
  - Research Site, Strathaven
  - Research Site, Sutton Coldfield
  - Research Site, Woodbridge
  - Research Site, Worthing

REFERENCES:
- [Derived] Halcox JP, Banegas JR, Roy C, Dallongeville J, De Backer G, Guallar E, Perk J, Hajage D, Henriksson KM, Borghi C. Prevalence and treatment of atherogenic dyslipidemia in the primary prevention of cardiovascular disease in Europe: EURIKA, a cross-sectional observational study. BMC Cardiovasc Disord. 2017 Jun 17;17(1):160. doi: 10.1186/s12872-017-0591-5. PMID 28623902
- [Derived] Borghi C, Rodriguez-Artalejo F, De Backer G, Dallongeville J, Medina J, Guallar E, Perk J, Banegas JR, Tubach F, Roy C, Halcox JP. The association between blood pressure and lipid levels in Europe: European Study on Cardiovascular Risk Prevention and Management in Usual Daily Practice. J Hypertens. 2016 Nov;34(11):2155-63. doi: 10.1097/HJH.0000000000001078. PMID 27512970
- [Derived] Borghi C, Tubach F, De Backer G, Dallongeville J, Guallar E, Medina J, Perk J, Roy C, Banegas JR, Rodriguez-Artalejo F, Halcox JP. Lack of control of hypertension in primary cardiovascular disease prevention in Europe: Results from the EURIKA study. Int J Cardiol. 2016 Sep 1;218:83-88. doi: 10.1016/j.ijcard.2016.05.044. Epub 2016 May 13. PMID 27232917
- [Derived] Halcox JP, Tubach F, Lopez-Garcia E, De Backer G, Borghi C, Dallongeville J, Guallar E, Medina J, Perk J, Sazova O, Sweet S, Roy C, Banegas JR, Rodriguez-Artalejo F. Low rates of both lipid-lowering therapy use and achievement of low-density lipoprotein cholesterol targets in individuals at high-risk for cardiovascular disease across Europe. PLoS One. 2015 Feb 18;10(2):e0115270. doi: 10.1371/journal.pone.0115270. eCollection 2015. PMID 25692692
- [Derived] Halcox JP, Roy C, Tubach F, Banegas JR, Dallongeville J, De Backer G, Guallar E, Sazova O, Medina J, Perk J, Steg PG, Rodriguez-Artalejo F, Borghi C. C-reactive protein levels in patients at cardiovascular risk: EURIKA study. BMC Cardiovasc Disord. 2014 Feb 24;14:25. doi: 10.1186/1471-2261-14-25. PMID 24564178
- [Derived] Halcox JP, Tubach F, Sazova O, Sweet S, Medina J; EURIKA steering committee. Reclassification of European patients' cardiovascular risk using the updated Systematic Coronary Risk Evaluation algorithm. Eur J Prev Cardiol. 2015 Feb;22(2):200-2. doi: 10.1177/2047487313507680. Epub 2013 Oct 3. PMID 24092875
- [Derived] Schmieder RE, Goebel M, Bramlage P. Barriers to cardiovascular risk prevention and management in Germany--an analysis of the EURIKA study. Vasc Health Risk Manag. 2012;8:177-86. doi: 10.2147/VHRM.S29915. Epub 2012 Mar 15. PMID 22536072
- [Derived] Dallongeville J, Banegas JR, Tubach F, Guallar E, Borghi C, De Backer G, Halcox JP, Masso-Gonzalez EL, Perk J, Sazova O, Steg PG, Artalejo FR; EURIKA Investigators. Survey of physicians' practices in the control of cardiovascular risk factors: the EURIKA study. Eur J Prev Cardiol. 2012 Jun;19(3):541-50. doi: 10.1177/1741826711407705. Epub 2011 Apr 18. PMID 21502280
- [Derived] Rodriguez-Artalejo F, Guallar E, Borghi C, Dallongeville J, De Backer G, Halcox JP, Hernandez-Vecino R, Jimenez FJ, Masso-Gonzalez EL, Perk J, Steg PG, Banegas JR; EURIKA Investigators. Rationale and methods of the European Study on Cardiovascular Risk Prevention and Management in Daily Practice (EURIKA). BMC Public Health. 2010 Jun 30;10:382. doi: 10.1186/1471-2458-10-382. PMID 20591142